CLINICAL TRIAL: NCT05485246
Title: Advanced Multimodal Anesthesia Care for Patients Undergoing Oro-maxillofacial Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-F(I)-20210211
Record Dates: First submitted 2022-05-15; First posted 2022-08-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-12

CONDITIONS: Orthognathic Surgery
Keywords: orthognathic surgery; anesthesia; prospective analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to develop from enhanced multimodal anesthesia care to verify and optimize ERAS strategies for orthognathic surgery. If the elements of anesthesia care can be accurately controlled, the harmful pressure factors caused by surgery can be minimized and the patients undergoing facial surgery can be improved.

DETAILED DESCRIPTION:
Orthognathic surgery (Orthognathic surgery) is currently one of the most commonly performed surgical items in oral and maxillofacial surgery because it corrects facial deformities, improves teeth chewing and face glowing. In general, the kind of operations are performed under nasotracheal intubating general anesthesia.

Due to the patients were required for motionless, low pressure, controlled ventilation, and adequate analgesia during anesthesia undergoing orthognathic surgery, advanced multimodal anesthesia care developing to the Enhanced Recovery After surgery (ERAS) should be conducted under patient safety. The ERAS concept emphasizes the importance of clinical multidisciplinary teamwork cooperation including of oro-surgeon, anesthesiologist, operating and post-anesthesia care nurses. The core elements of ERAS lies in the management of the entire peri-operative period of anesthesia. In clinical practice, focus on entire anesthesia care during the operation includes of precise anesthesia depth, adequate muscle relaxation, multiple modes of pain controlled and adequate analgesia, stable body temperature maintenance, use of goal-oriented infusion therapy, early extubation, and prevention of postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* America society anesthesiologist classification class I to III patients undergoing oro-maxillo-facial surgery
* unlimited mouth opening
* nasotracheal intubation general anesthesia for at least 120 minutes.

Exclusion criteria:

* patients with arthritis with limited mouth opening
* diabetes with insulin treatment
* essential hypertension without controlled
* past history of malignant hyperthermia or personal or family history
* persistent liver dysfunction
* chronic renal insufficiency
* body mass index ≧35 kg/m2.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without obviously systemic diseases who presentation of abnormal oro-maxillofacial anatomy needs to be corrected.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
permitted hypotension during surgery with adequate depth of anesthesia and cardiac output | intraoperative 2-6 hours
  to decrease intra-operative bleeding as patient undergoing oromaxillofacial surgery, intentional hypotension is allowed. however, adequate depth of anesthesia, proper cardiac output, respiratory parameters, temperatures should be monitored
consumption of inhaled and intravenous anesthetics | intraoperative 2-6 hours
  to maintain adequate depth of anesthesia during intentional hypotension, consumptions of inhaled and intravenous anesthetics are calculated

SECONDARY OUTCOMES:
time to successfully extubate the nasotracheal tube after anesthesia | from the end of surgery to the post-anesthesia care, assessed up to one hour
  early extubation allowable
safely discharged from post-anesthesia care unit (postoperative recovery room) | 2 hours
  as calculating the time from patient is delivered to postoperative recovery room to be safely discharged from recovery room by using the aldrete scores (activities level, respiration, circulation, conscious level, oxygenation) full back to pre-operative level or ten scores.
side effects and adverse events | intraoperative and postoperative stages, assessed up to 48 hours
  records any abnormal surgical or anesthesia related findings during this admission

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-I Cheng, Phd, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan